CLINICAL TRIAL: NCT05323383
Title: The Effects and Mechanisms of Brief Training in Mindfulness Meditation and Hypnosis for Pain Management, Relative to an Inert Control
Brief Title: The Effects and Mechanisms of Brief Mindfulness Meditation and Hypnosis for Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/HE000347
Record Dates: First submitted 2022-03-15; First posted 2022-04-12 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-08

CONDITIONS: Pain; Chronic Pain
MeSH Terms: conditions — Pain; Chronic Pain | interventions — Mindfulness; Hypnosis

STUDY DESIGN:
Intervention Model Description: Single-blind, three-arm, parallel-group randomized design
Who Masked: Outcomes Assessor
Masking Description: Outcomes are assessed remotely via Qualtrics, thus the outcome "assessor" is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness meditation (Experimental): Participants in the mindfulness meditation condition will practice one, 20-minute breath and body focused meditation.
  Interventions: Behavioral: Mindfulness Meditation
- Self-Hypnosis (Active Comparator): Participants in self-hypnosis will practice one, 20-minute audio-guided hypnosis session with suggestions tailored towards enhancing positive affect and fostering decentering.
  Interventions: Behavioral: Self-hypnosis
- Control (Other): Participants in the attention control condition will listen to a 20-minute natural history recording.
  Interventions: Other: Attention Control

INTERVENTIONS:
Behavioral: Mindfulness Meditation — Participants in the mindfulness meditation condition will listen to a 20minute guided mindfulness meditation practice that holds the breath and body as the object of meditation.
  Arms: Mindfulness meditation
Behavioral: Self-hypnosis — Participants in self-hypnosis will listen to a 20-minute audio-guided hypnosis practice with an induction phase, followed by suggestions tailored towards shifts in affect and decentering, and then a re-alerting with post-hypnotic suggestions phase.
  Arms: Self-Hypnosis
Other: Attention Control — Control participants will listen to a 20-minute natural history recording which was chosen as past research has found that individuals who listen to it report this to be a neutral, but relaxing passage, and it has been used as an effective control condition in previous research.
  Arms: Control

SUMMARY:
The aim of this study is to determine the effects and mechanisms of 1 x 20-min training in mindfulness meditation and self-hypnosis relative to an inert control. Participants will be randomly assigned to condition. The dual primary outcomes will be pre- to post-training changes in current pain intensity and pain unpleasantness. The active treatments are hypothesized to produce greater reductions in pain outcomes than the control. It is also hypothesized that change in mindfulness will be a mediator specific to mindfulness meditation, while change in affect and decentering will be mediators of the hypnosis condition. Moderators of response will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age;
* Experience chronic or recurrent pain;
* Have access to a computer, phone or tablet with internet capability; and
* Be able to read and understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Current pain intensity | Change from pre- (Time 1; start of survey) to post-20-min training (Time 2; following completion of the one, 20-min training)
  Numerical rating scale ranging from 0-10
Current pain unpleasantness | Change from pre- (Time 1; start of survey) to post-20-min training (Time 2; following completion of the one, 20-min training)
  Numerical rating scale ranging from 0-10

SECONDARY OUTCOMES:
Mechanism: Mindfulness | Change from pre- (Time 1; start of survey) to post-20-min training (Time 2; following completion of the one, 20-min training)
  State Mindfulness Scale with items ranging from 1-5
Mechanism: Positive Affect | Change from pre- (Time 1; start of survey) to post-20-min training (Time 2; following completion of the one, 20-min training)
  PANAS-X
Mechanism: Decentering | Change from pre- (Time 1; start of survey) to post-20-min training (Time 2; following completion of the one, 20-min training)
  State decentering MpoD-s

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Queensland, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided
The dataset generated and analysed during the current study will be available from the corresponding author on reasonable request once published. The data will not be not publicly available due to ethical restrictions.